CLINICAL TRIAL: NCT05917366
Title: The Effectiveness of Manipulation in Combination With Exercise for Patients With Coccydynia: A Randomized Controlled Trial
Brief Title: Effect of Manipulation on Coccydynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KaratayManipulation
Record Dates: First submitted 2023-06-06; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Coccyx Disorder; Pelvic Floor; Weak; Stretch
MeSH Terms: conditions — Asthenia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coccyx Manipulation (Experimental): Manual therapy sessions, in addition to the exercise group, were performed once a week for four weeks.
  Interventions: Other: Exercises; Other: Coccyx Manipulation
- Exercises (Active Comparator): A total of 4 sessions were applied, 3 times a week.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Stretching exercise for the piriformis and iliopsoas muscles. strengthening exercises for pelvic floor muscles
Other: Coccyx Manipulation — Application of manipulation to relax the levetor ani muscle
  Arms: Coccyx Manipulation

SUMMARY:
The aim of this study was to investigate the efficacy of manipulation combined with exercise as a treatment for patients with coccydynia.

DETAILED DESCRIPTION:
Subject: Coccydynia is a painful condition characterized by inflammation and discomfort in the coccyx region, commonly known as the tailbone. It can significantly affect an individual's quality of life by impairing their ability to sit, stand, or engage in daily activities. Various treatment approaches have been explored to alleviate the symptoms of coccydynia, including manipulation techniques and exercise interventions. However, to date, there is a scarcity of research investigating the combined effects of manipulation and exercise for patients with coccydynia.

Purpose: The purpose of this study is to evaluate the efficacy of combining manipulation techniques with exercise interventions for patients diagnosed with coccydynia, a painful condition affecting the coccyx region. Despite the debilitating impact of coccydynia on daily activities and quality of life, there is a limited understanding of the optimal treatment approach for this condition. This study aims to address this knowledge gap by investigating the potential benefits of combining manipulation and exercise in managing coccydynia.

ELIGIBILITY:
Inclusion Criteria:

* chronic (3 months) coccydynia
* age over 25 and under 60 years
* no ongoing antidepressant treatment
* no medicolegal litigation or occupational-accident etiology

Exclusion Criteria:

* undergoing an operation aimed at the anal area
* those with additional diseases such as radiculopathy etc.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-07-16 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain at 4 weeks and 6 months | Baseline measurement before the treatment programs begin (pre-intervention), post-intervention at week 4, and 6 months follow-up
  A visual analog scale (VAS) numbered 0-10 will be used in the assessment of pain.
Change from baseline in Paris questionnaire at 4 weeks and 6 months | Baseline measurement before the treatment programs begin (pre-intervention), post-intervention at week 4, and 6 months follow-up
  Coccydynia-related symptoms were recorded using the Paris questionnaire, ranging from 0 (no symptoms) to 10 (maximum symptoms). The Paris questionnaire is a specific assessment tool designed to evaluate symptoms and functional limitations related to coccydynia, a condition characterized by pain in the coccyx region. The questionnaire consists of a series of questions that inquire about the severity and impact of coccyx pain on various activities and daily life.
Change from baseline in The Oswestry Disability Index at 4 weeks and 6 months | Baseline measurement before the treatment programs begin (pre-intervention), post-intervention at week 4, and 6 months follow-up
  The Oswestry Disability Index consists of ten sections, each addressing a different aspect of functional ability, including pain intensity, lifting, ability to walk, ability to sit, ability to stand, sleep quality, ability to socialize, ability to travel, ability to perform self-care tasks, and ability to perform household tasks. Each section contains multiple statements, and the individual rates their level of disability on a scale of 0 to 5, with higher scores indicating greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Sönmez ÜNÜVAR, Principal Investigator — KTO KARATAY UNIVERSTESI
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No